CLINICAL TRIAL: NCT03149796
Title: The Effect of Tocilizumab (Anti-interleukin-6) Treatment on microRNA Expression and Adipokine Levels in Rheumatoid Arthritis Patients
Brief Title: Tocilizumab Effect on microRNA Expression and Adipokine Levels in Rheumatoid Arthritis Patients
Status: Completed | Type: Observational
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Devy Zissman, head of rheumatology department, Carmel Medical Center
Other Study IDs: CMC-11-0018-CTIL
Record Dates: First submitted 2017-05-10; First posted 2017-05-11 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — periferal blood and serum

GROUPS / COHORTS (2):
- RA patients: designated to be treated with tocilizumab and followed in rheumatology clinics.
  Laboratory blood tests will be collected and analyzed
  Interventions: Other: laboratory blood tests
- healthy controls: control Laboratory blood tests will be collected and analyzed
  Interventions: Other: laboratory blood tests

INTERVENTIONS:
Other: laboratory blood tests — Serum concentrations of leptin, adiponectin, resistin, interleukin-6 and high sensitivity C reactive protein were measured by ELISA in both study groups

SUMMARY:
The investigators propose to identify changes in cytokines like adipocytokines and microRNA (miR) expression (for example miR-9, miR-16, miR-125, miR-132, miR-146a, miR-150, miR-155, miR-181 and miR-223) in peripheral blood leukocytes and in serum samples obtained from rheumatoid arthritis (RA) patients before and after tocilizumab treatment. The results obtained will be compared to gender- and age-matched healthy controls, and will help the investigators define one or more miRNAs as biomarkers for treatment effectiveness.

Methods The investigators will obtain blood samples from 60 RA patients treated with tocilizumab, according to the local clinical guidelines. Blood samples will be collected before treatment, as well as one and four months following tocilizumab treatment. The blood samples will initially undergo microarray analysis and then the results will be confirmed for specific miRNAs by quantitative real-time PCR (qPCR). The serum level of the tested cytokines, like adipokines, will be measured using ELISA methods. The changes in cytokines level and miRNAs expression, either up-regulation or down-regulation, during tocilizumab therapy will be correlated to the severity of the disease and to specific demographic and medical data. The results obtained will be compared to 60 healthy controls gender- and age-matched

DETAILED DESCRIPTION:
The aim of the study is to investigate the effects of tocilizumab on the expression of biomarkers like adipocytokines and miRNAs in peripheral blood leukocytes and in serum samples obtained from rheumatoid arthritis patients. Candidate miRNAs that are likely to be quantitated are for example miR-9, 16, 125, 132, 146a, 150, 155, 181 and, 223. The results obtained will help the investigators determine if cytokines and miRNAs expression can be used as a novel biomarker for the determination of the effectiveness of tocilizumab treatment.

The study is designed as a prospective study investigating the effect of tocilizumab on the expression of cytokines and miRNA in rheumatoid arthritis patients. Sixty rheumatoid arthritis patients designated to be treated with tocilizumab and followed in rheumatology clinics.

After receiving informed consent, three blood samples of 5cc blood each will be drawn: the first - before tocilizumab treatment to set the basal level of expression in untreated patients, the second and third samples will be taken one month and four months after initiation of tocilizumab treatment. The investigators will use selected samples (from 5 patients) to perform microarray analysis for miRNAs expression, and based on the results, we will confirm the expression of specific miRNAs by quantitative real-time PCR (qPCR). Based on current knowledge, the investigators expect that miR-9, 16, 125, 132, 146a, 150, 155, 181 and, 223 will show significant changes in expression upon tocilizumab treatment. Cytokines levels are measured using ELISA tests for each individual biomarker. The changes in cytokines and miRNAs expression, either up-regulation or down-regulation, will be correlated to the severity of the disease and to the clinical effect of tocilizumab. Information regarding disease duration, activity as measured by disease activity score, concomitant treatment and serology status will be collected. Also demographic characteristics - age, sex and smoking status will be recorded. The results will be compared to 60 healthy controls gender- and age matched, without any rheumatic, inflammatory or malignant disorders

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfilling the 2010 Rheumatoid Arthritis Classification criteria.
* Patients designated to tocilizumab treatment
* Age above 18 years old
* Signed informed concern
* Ability to read and write in Hebrew

Exclusion Criteria:

* Patients with other rheumatic diseases
* Patients with other inflammatory diseases
* Patients with malignancies

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: RA patients treated with tocilizumab, according to the local clinical guidelines
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2011-03-23 (Actual); Primary Completion 2013-05-01 (Actual); Study Completion 2013-05-01 (Actual)

PRIMARY OUTCOMES:
expression of biomarkers like adipocytokines and miRNAs | four months
  expression of biomarkers like adipocytokines and miRNAs in peripheral blood leukocytes and in serum samples obtained from RA patients. Candidate miRNAs that are likely to be quantitated are for example miR-9, 16, 125, 132, 146a, 150, 155, 181 and, 223

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Barton A, Worthington J. Genetic susceptibility to rheumatoid arthritis: an emerging picture. Arthritis Rheum. 2009 Oct 15;61(10):1441-6. doi: 10.1002/art.24672. No abstract available. PMID 19790122
- [Background] Symmons D, Harrison B. Early inflammatory polyarthritis: results from the norfolk arthritis register with a review of the literature. I. Risk factors for the development of inflammatory polyarthritis and rheumatoid arthritis. Rheumatology (Oxford). 2000 Aug;39(8):835-43. doi: 10.1093/rheumatology/39.8.835. No abstract available. PMID 10952736
- [Background] Lard LR, Visser H, Speyer I, vander Horst-Bruinsma IE, Zwinderman AH, Breedveld FC, Hazes JM. Early versus delayed treatment in patients with recent-onset rheumatoid arthritis: comparison of two cohorts who received different treatment strategies. Am J Med. 2001 Oct 15;111(6):446-51. doi: 10.1016/s0002-9343(01)00872-5. PMID 11690569
- [Background] Firestein GS. Evolving concepts of rheumatoid arthritis. Nature. 2003 May 15;423(6937):356-61. doi: 10.1038/nature01661. PMID 12748655
- [Background] Redlich K, Hayer S, Ricci R, David JP, Tohidast-Akrad M, Kollias G, Steiner G, Smolen JS, Wagner EF, Schett G. Osteoclasts are essential for TNF-alpha-mediated joint destruction. J Clin Invest. 2002 Nov;110(10):1419-27. doi: 10.1172/JCI15582. PMID 12438440
- [Background] Feldmann M, Brennan FM, Maini RN. Role of cytokines in rheumatoid arthritis. Annu Rev Immunol. 1996;14:397-440. doi: 10.1146/annurev.immunol.14.1.397. PMID 8717520
- [Background] Kotake S, Udagawa N, Takahashi N, Matsuzaki K, Itoh K, Ishiyama S, Saito S, Inoue K, Kamatani N, Gillespie MT, Martin TJ, Suda T. IL-17 in synovial fluids from patients with rheumatoid arthritis is a potent stimulator of osteoclastogenesis. J Clin Invest. 1999 May;103(9):1345-52. doi: 10.1172/JCI5703. PMID 10225978
- [Background] Dayer JM, Choy E. Therapeutic targets in rheumatoid arthritis: the interleukin-6 receptor. Rheumatology (Oxford). 2010 Jan;49(1):15-24. doi: 10.1093/rheumatology/kep329. Epub 2009 Oct 23. PMID 19854855
- [Background] Eastgate JA, Symons JA, Wood NC, Grinlinton FM, di Giovine FS, Duff GW. Correlation of plasma interleukin 1 levels with disease activity in rheumatoid arthritis. Lancet. 1988 Sep 24;2(8613):706-9. doi: 10.1016/s0140-6736(88)90185-7. PMID 2901567
- [Background] van Leeuwen MA, Westra J, Limburg PC, van Riel PL, van Rijswijk MH. Clinical significance of interleukin-6 measurement in early rheumatoid arthritis: relation with laboratory and clinical variables and radiological progression in a three year prospective study. Ann Rheum Dis. 1995 Aug;54(8):674-7. doi: 10.1136/ard.54.8.674. PMID 7677445
- [Background] Taganov KD, Boldin MP, Baltimore D. MicroRNAs and immunity: tiny players in a big field. Immunity. 2007 Feb;26(2):133-7. doi: 10.1016/j.immuni.2007.02.005. PMID 17307699
- [Background] Shi XB, Tepper CG, deVere White RW. Cancerous miRNAs and their regulation. Cell Cycle. 2008 Jun 1;7(11):1529-38. doi: 10.4161/cc.7.11.5977. Epub 2008 Mar 20. PMID 18469525
- [Background] Williams AE, Perry MM, Moschos SA, Larner-Svensson HM, Lindsay MA. Role of miRNA-146a in the regulation of the innate immune response and cancer. Biochem Soc Trans. 2008 Dec;36(Pt 6):1211-5. doi: 10.1042/BST0361211. PMID 19021527
- [Background] Baltimore D, Boldin MP, O'Connell RM, Rao DS, Taganov KD. MicroRNAs: new regulators of immune cell development and function. Nat Immunol. 2008 Aug;9(8):839-45. doi: 10.1038/ni.f.209. PMID 18645592
- [Background] O'Connell RM, Taganov KD, Boldin MP, Cheng G, Baltimore D. MicroRNA-155 is induced during the macrophage inflammatory response. Proc Natl Acad Sci U S A. 2007 Jan 30;104(5):1604-9. doi: 10.1073/pnas.0610731104. Epub 2007 Jan 22. PMID 17242365
- [Background] Taganov KD, Boldin MP, Chang KJ, Baltimore D. NF-kappaB-dependent induction of microRNA miR-146, an inhibitor targeted to signaling proteins of innate immune responses. Proc Natl Acad Sci U S A. 2006 Aug 15;103(33):12481-6. doi: 10.1073/pnas.0605298103. Epub 2006 Aug 2. PMID 16885212
- [Background] Luo X, Tsai LM, Shen N, Yu D. Evidence for microRNA-mediated regulation in rheumatic diseases. Ann Rheum Dis. 2010 Jan;69 Suppl 1:i30-36. doi: 10.1136/ard.2009.117218. PMID 19995741
- [Background] Pauley KM, Satoh M, Chan AL, Bubb MR, Reeves WH, Chan EK. Upregulated miR-146a expression in peripheral blood mononuclear cells from rheumatoid arthritis patients. Arthritis Res Ther. 2008;10(4):R101. doi: 10.1186/ar2493. Epub 2008 Aug 29. PMID 18759964
- [Background] Meng F, Henson R, Wehbe-Janek H, Smith H, Ueno Y, Patel T. The MicroRNA let-7a modulates interleukin-6-dependent STAT-3 survival signaling in malignant human cholangiocytes. J Biol Chem. 2007 Mar 16;282(11):8256-64. doi: 10.1074/jbc.M607712200. Epub 2007 Jan 12. PMID 17220301
- [Background] Trenkmann M, Brock M, Ospelt C, Gay S. Epigenetics in rheumatoid arthritis. Clin Rev Allergy Immunol. 2010 Aug;39(1):10-9. doi: 10.1007/s12016-009-8166-6. PMID 19707891
- [Background] Lotvall J, Valadi H. Cell to cell signalling via exosomes through esRNA. Cell Adh Migr. 2007 Jul-Sep;1(3):156-8. doi: 10.4161/cam.1.3.5114. Epub 2007 Jul 4. PMID 19262134
- [Background] Rho YH, Solus J, Sokka T, Oeser A, Chung CP, Gebretsadik T, Shintani A, Pincus T, Stein CM. Adipocytokines are associated with radiographic joint damage in rheumatoid arthritis. Arthritis Rheum. 2009 Jul;60(7):1906-14. doi: 10.1002/art.24626. PMID 19565493